CLINICAL TRIAL: NCT02458222
Title: Efficacy of Language Games as Therapy for Post Stroke Aphasia
Acronym: AphasiaGame
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RG_14-300
Record Dates: First submitted 2015-05-01; First posted 2015-06-01 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Stroke; Aphasia
MeSH Terms: conditions — Stroke; Aphasia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- game therapy then standard therapy (Experimental): participants will take part in language game therapy followed by standard aphasia therapy
  Interventions: Other: language game therapy; Other: standard therapy
- standard therapy then game therapy (Experimental): participants will have standard aphasia therapy first then will take part in language game therapy
  Interventions: Other: language game therapy; Other: standard therapy

INTERVENTIONS:
Other: language game therapy — participants will take part in game therapy
Other: standard therapy — usual clinical care

SUMMARY:
Aphasia is a language impairment experienced by about one third of stroke patients. This often devastating condition is treated by speech and language therapists (SLTs). There is evidence that language games delivered at the right intensity are an efficacious means of improving communication for people with post stroke aphasia. However, it is unclear which mechanism of language facilitation used in a game works best. This study will provide evidence for the "active ingredient" of a game, together with measures of efficacy, feasibility and enjoyment compared to standard aphasia therapy.

DETAILED DESCRIPTION:
Aphasia is a language impairment experienced by about one third of stroke patients. This often devastating condition is treated by speech and language therapists (SLTs). There is evidence that language games delivered at the right intensity are an efficacious means of improving communication for people with post stroke aphasia. However, it is unclear which mechanism of language facilitation used in a game works best. This study will provide evidence for the "active ingredient" of a game, together with measures of efficacy, feasibility and enjoyment compared to standard aphasia therapy.

Participants with moderate-severe difficulties will play picture naming games, involving self-cuing using gesture and circumlocution. Those with mild difficulties will play story-telling games, using similar self-cuing techniques. Change in language performance will be measured and compared to that achieved by the same participants following an episode of standard aphasia therapy from their local SLT (i.e. normal care).

This study will build on a growing evidence base for the efficacy of therapeutic language games in post stroke aphasia. In today's resource-constrained National Health Service, SLTs are continually searching for cost-effective, innovative ways of delivering therapy. Language games based on sound neuro-scientific principles have the potential to deliver improvements in functional communication by means of an enjoyable and motivating activity, and moreover can be done cost effectively. Improvements have been demonstrated from the acute through to the chronic stage of stroke. A number of factors are said to contribute to the outcomes achieved: intensity of training, behavioural relevance and focussed use of capacities. This study intends to explore in more depth some of the specific behaviours that can occur spontaneously or than can be prompted to facilitate language. The aim is to uncover the "active ingredient", and thereby ensure that participants can benefit maximally from therapeutic language games.

This study will contribute to the search for cost effective treatment for post-stroke aphasia, which offers ease and flexibility of delivery, is enjoyable and motivating for patients, and works.

ELIGIBILITY:
Inclusion Criteria:

* Adults who have suffered a stroke a minimum of 2 months prior to commencement of the intervention. They will present with expressive aphasia, with relatively preserved language comprehension. They will have been fully fluent in English before the stroke.

Exclusion Criteria:

* Severe perceptual or cognitive deficits. History of other neurological, psychiatric or neurodegenerative disease impairing language or communicative ability. Severe visual agnosia. Severe limb apraxia. Severe dysarthria. Drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Aphasia Test (Swinburn et al 2004) | Assessment carried out prior to commencement of language game therapy, and immediately after language game therapy, 10 week interval. Assessment also carried out prior to and immediately after standard therapy, approx 12 week interval.
  Measures of language performance taken as designated in the various sub-tests, and comparisons of improvement in those measures after game therapy and after standard therapy. These will measure the general efficacy of the intervention.
Communication Outcomes After Stroke Scale (Long et al, 2008) | Assessment carried out prior to commencement of language game therapy, and immediately after language game therapy, 10 week interval. Assessment also carried out prior to and immediately after standard therapy, approx 12 week interval.
  Measures of participants' subjective views of communicative abilities taken as designated by the test, and comparisons of improvement in those measures after game therapy and after standard therapy. These will measure the impact of therapy on general functional communication.
Picture naming of words targeted in game therapy | Assessment carried out prior to commencement of language game therapy, and immediately after language game therapy, 10 week interval. Assessment also carried out prior to and immediately after standard therapy, approx 12 week interval.
  Confrontational picture naming of 180 words targeted in game therapy- points awarded for correct naming, and comparisons of improvement in those measures after game therapy and after standard therapy. These will measure therapy effects for the items that are specifically treated based on single word production.
Picture description of words targeted in game therapy | Assessment carried out prior to commencement of language game therapy, and immediately after language game therapy, 10 week interval. Assessment also carried out prior to and immediately after standard therapy, approx 12 week interval.
  Measures of improvement in connected speech using method from Comprehensive Aphasia Test. Comparison of improvement following game therapy and following standard therapy. These will measure the ability of participants to use targeted words, but in a functional communication context -- i.e. producing phrases and sentences to describe a scene.

SECONDARY OUTCOMES:
Picture naming of words targeted in game therapy to ascertain effects of different facilitatory techniques - multiple baseline measure | Assessment carried out immediately after game 1 and game 2, at 4 weeks and 7 weeks.
  Confrontational picture naming of 180 words targeted in game therapy- points awarded for correct naming, and comparisons of improvement in those measures after each type of language game.
Picture description of words targeted in game therapy to ascertain effects of different facilitatory techniques - multiple baseline measure | Assessment carried out immediately after game 1 and game 2, at 4 weeks and 7 weeks.
  Measures of improvement in connected speech using method from Comprehensive Aphasia Test. Comparison of improvement following each type of language game.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Jennings, PhD, Study Chair — University of Birmingham
Locations (1):
- Moor Green Out-Patient Brain Injury Service, Birmingham, West Midlands, United Kingdom